CLINICAL TRIAL: NCT04695613
Title: Amino Acids Versus Magnesium Sulphate Infusion in Controlling Postoperative Shivering
Brief Title: Shivering Control After Percutaneous Nephrolithotomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Makram Soliman, lecturer of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17300539
Record Dates: First submitted 2021-01-03; First posted 2021-01-05 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Shivering Control
MeSH Terms: interventions — Amino Acids; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aminoacid group (Active Comparator): patients received an IV amino acid infusion 150 ml/kg/hr starting just before and during anesthesia
  Interventions: Drug: Aminoacid
- magnesium sulfate group (Active Comparator): patients received an IV magnesium sulphate bolus and infusion 40 mg/kg starting just before and during anesthesia
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Aminoacid — amino acid infusion 150 ml/kg/hr starting preoperative
  Arms: aminoacid group
Drug: Magnesium sulfate — magnesium sulphate bolus and infusion 60 mg/kg starting preoperative
  Arms: magnesium sulfate group

SUMMARY:
Aim of the study is comparing the effect of amino acid versus magnesium sulfate infusion on postoperative shivering in patients undergoing elective percutaneous nephrolithotomy surgery under general anesthesia.

DETAILED DESCRIPTION:
A written informed consent was taken from the patients. Patients were assigned randomly to two groups (40 subjects each) to be anesthetized and infused with either an iv amino acid starting just before and during anesthesia (group A) or an iv magnesium sulphate starting just before and during anesthesia (group M) in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II who were listed for elective percutaneous nephrolithotomy PCNL surgery under general anesthesia.

Exclusion Criteria:

* Hepatic inefficiency
* Renal inefficiency
* Spinal anesthesia because of a different mechanism of hypothermia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Postoperative shivering grade | 2 hours postoperative
  "grading of shivering," in which shivering degree was assessed as 1 of 5 levels (0, 1, 2, 3, and 4), grade 0 lack of shivering, grade 1 slight shivering (inconsiderable yet apparent peripheral vasoconstriction), grade 2 medium level shivering (muscular activity in one muscle group only) grade 3 severe shivering (muscular activity in more than one muscle group without generalized shivering) and grade 4 generalized shivering.

SECONDARY OUTCOMES:
Shivering frequency | 2 hours postoperative
  Number of shivering episodes in postoperative period
Blood loss volume | 2 hours postoperative
  Assessing blood loss in surgical drains postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt